CLINICAL TRIAL: NCT01326949
Title: Transjugular Intrahepatic Portosystemic Shunt Versus Endoscopic Treatment Combined With Propranolol for Prevention of Variceal Rebleeding in Cirrhotic Patients With Portal Vein Thrombosis: A Randomized Controlled Trial
Brief Title: Transjugular Intrahepatic Portosystemic Shunt (TIPS) for Prevention of Variceal Rebleeding in Cirrhotic Patients With Portal Vein Thrombosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Guohong Han, Head of Department of Digestive Interventional Radiology, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1PVT-TIPS
Record Dates: First submitted 2011-03-29; First posted 2011-03-31 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Decompensated Cirrhosis; Portal Vein Thrombosis; Bleeding Varices
MeSH Terms: interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ET+NSBB (Active Comparator): Endoscopic treatment(ET)- Endoscopic variceal ligation (EVL)
  Non-selective beta blocker(NSBB)-Propranolol.
  Anticoagulation(AT)- Heparin followed by warfarin.
  Interventions: Procedure: ET+NSBB
- TIPS (Active Comparator): Transjugular intrahepatic portosystemic shunt(TIPS)- TIPS.
  Interventions: Procedure: Transjugular intrahepatic portosystemic shunt (TIPS)

INTERVENTIONS:
Procedure: Transjugular intrahepatic portosystemic shunt (TIPS) — Transjugular intrahepatic portosystemic shunt(TIPS)- TIPS was performed in a conventional fashion or in combination of percutaneous transhepatic or transsplenic approach. Postoperatively, intravenous heparin (8,000-12,000 u/d) for five days, warfarin for six months were given.
  Arms: TIPS
Procedure: ET+NSBB — ET-Esophageal varices was treated by endoscopic variceal ligation (EVL). EVL was repeated at intervals of 1-2 weeks until the varices were obliterated or reduced to grade-I size.
  NSBB-Propranolol started at a dose of 20mg twice a day. The dose is adjusted to the maximal tolerated doses to heart rate (HR) of 55 bpm or to decrease the HR 25% from baseline.
  AT-A continuously intravenous infusion of unfractionated heparin followed by oral warfarin is employed. Initially, heparin is administered intravenously for 5 days. Subsequently, oral warfarin is prescribed at the dosage of 2.5 mg/d for 6 months or until complete portal vein recanalization and adjusted to maintain the INR at a target of 2.5 (range 2.0-3.0).
  Arms: ET+NSBB

SUMMARY:
Portal vein thrombosis (PVT) refers to an obstruction in the trunk of the portal vein. It can extend downstream to the portal branches, or upstream to the splenic and/or the mesenteric veins. The prevalence of PVT is 10-25% and incidence is about 16% in cirrhotic patients. Recent studies demonstrate that the presence of PVT is not only an independent predictor of failure to control active variceal bleeding and prevent variceal rebleeding, but also significantly associated with increased mortality in patients with liver cirrhosis.

However, in recent American Association of the Study of Liver Disease (AASLD) practice guidelines and Baveno V consensus, no treatment strategies in cirrhotic patients with PVT was clearly recommended due to the absence of randomized controlled trials.

DETAILED DESCRIPTION:
Usually, cirrhotic patients with PVT are submitted to variceal rebleeding prophylaxis with endoscopic band ligation combined with non-selective beta-blockers and, when necessary, the anticoagulation is started after the varices eradication.

TIPS is just regarded as the second-line therapy for the secondary prophylaxis of variceal bleeding in cirrhotic patients. However, this indication might be changed in the setting of PVT. Indeed, the risk to benefit ratio of TIPS in cirrhotic patients with PVT for the prevention of recurrent variceal bleeding has never been evaluated.

The aim of this study is to compare the efficacy and safety of TIPS and endoscopic band ligation + propranolol in decompensated cirrhosis patients with PVT and a history of variceal bleeding in the past 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Liver cirrhosis
* Portal vein thrombosis (degree of vessel obstruction > 50%)
* History of variceal hemorrhage in the past 6 weeks (recent variceal bleeding has been controlled for at least 120 hours)

Exclusion Criteria:

* Uncontrolled active variceal bleeding
* Fibrotic cord of the portal vein
* Prior history of TIPS placement or shunt surgery or endoscopic ban ligation +NSBB
* Concomitant renal insufficiency
* Severe cardiopulmonary diseases
* Uncontrolled systemic infection or sepsis
* Malignancy or other serious medical illness which may reduce the life expectancy
* Contraindications for propranolol, such as asthma, insulin-dependent diabetes (with episodes of hypoglycemia), and peripheral vascular disease
* Contraindications for heparin or warfarin
* Contraindications for TIPS

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with variceal rebleeding | 4 years
  Variceal rebleeding is the primary endpoint of this study. Cumulative variceal rebleeding rate is compared between the two groups.

SECONDARY OUTCOMES:
Number of death | 4 years
  Death is a secondary endpoint of this study. Cumulative survival rate is compared between the two groups.
Number of participants achieving portal vein recanalization | 4 years
  Portal vein recanalization is a secondary endpoint of this study. Recanalization rate of thrombosed portal vein is compared between the two groups.
Changes of degree of PVT in patients without portal vein recanalization | 4 years
  We also observed changes of degree of portal vein thrombosis in patients without portal vein recanalization.
Number of complications | 4 years
  Complications include:
  TIPS-related complications: procedural complications, shunt dysfunction and hepatic encephalopathy.
  Complications related to endoscopic and drug treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Guohong Han, Principal Investigator — Xijing Hospital of Digestive Diseases, Fourth Military Medical University
Locations (1):
- Xijing Hospital of Digestive Diseases, Fourth Military Medical University, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Han G, Qi X, He C, Yin Z, Wang J, Xia J, Yang Z, Bai M, Meng X, Niu J, Wu K, Fan D. Transjugular intrahepatic portosystemic shunt for portal vein thrombosis with symptomatic portal hypertension in liver cirrhosis. J Hepatol. 2011 Jan;54(1):78-88. doi: 10.1016/j.jhep.2010.06.029. Epub 2010 Aug 27. PMID 20932597
- [Derived] Simonetti RG, Perricone G, Robbins HL, Battula NR, Weickert MO, Sutton R, Khan S. Portosystemic shunts versus endoscopic intervention with or without medical treatment for prevention of rebleeding in people with cirrhosis. Cochrane Database Syst Rev. 2020 Oct 22;10(10):CD000553. doi: 10.1002/14651858.CD000553.pub3. PMID 33089892
- [Derived] Lv Y, Qi X, He C, Wang Z, Yin Z, Niu J, Guo W, Bai W, Zhang H, Xie H, Yao L, Wang J, Li T, Wang Q, Chen H, Liu H, Wang E, Xia D, Luo B, Li X, Yuan J, Han N, Zhu Y, Xia J, Cai H, Yang Z, Wu K, Fan D, Han G; PVT-TIPS Study Group.. Covered TIPS versus endoscopic band ligation plus propranolol for the prevention of variceal rebleeding in cirrhotic patients with portal vein thrombosis: a randomised controlled trial. Gut. 2018 Dec;67(12):2156-2168. doi: 10.1136/gutjnl-2017-314634. Epub 2017 Sep 28. PMID 28970291
- [Derived] Qi X, He C, Yin Z, Wang Z, Zhang H, Yao L, Wang J, Xia J, Cai H, Yang Z, Bai M, Guo W, Niu J, Wu K, Fan D, Han G; PVT-TIPS Study Group. Transjugular intrahepatic portosystemic shunt for the prevention of variceal rebleeding in cirrhotic patients with portal vein thrombosis: study protocol for a randomised controlled trial. BMJ Open. 2013 Jul 11;3(7):e003370. doi: 10.1136/bmjopen-2013-003370. Print 2013. PMID 23847271